CLINICAL TRIAL: NCT00384475
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study Using the Environmental Exposure Chamber (EEC) to Assess the Onset of Action of Ciclesonide, Applied as a Nasal Spray (200 mcg, Once Daily), in the Treatment of Seasonal Allergic Rhinitis (SAR) in Patients 18 Years and Older
Brief Title: A Study of Ciclesonide Nasal Spray in Patients 18 Years and Older With Seasonal Allergic Rhinitis (BY9010/M1-413)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-413
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Rhinitis, Allergic, Seasonal; Hay Fever
Keywords: Seasonal Allergic Rhinitis; Ciclesonide; Hay Fever; SAR
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

INTERVENTIONS:
Drug: Ciclesonide Nasal Spray

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of ciclesonide nasal spray as compared with placebo (inactive substance) nasal spray in relieving symptoms of seasonal allergic rhinitis caused by pollen. Ciclesonide will be administered once during the exposure to ragweed pollen in a controlled environment. The study duration consists of a baseline period (up to 5 days) and a treatment period (1 day). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* General good health
* History of SAR to short ragweed pollen for 2 years immediately preceding the study
* Demonstrated sensitivity to short ragweed known to induce SAR through a standard skin prick test

Main Exclusion Criteria:

* Clinically significant physical finding of nasal anatomical deformities causing greater than 50% obstruction, including but not limited to nasal polyps, septal defects, respiratory tract malformations, nasal trauma or surgery
* Known hypersensitivity to any corticosteroid
* History of a respiratory infection or disorder including but not limited to bronchitis, pneumonia, chronic sinusitis, influenza or SARS (severe acute respiratory syndrome) within 14 days preceding the Screening Visit
* History of alcohol or drug abuse within 2 years preceding the Screening Visit
* Active asthma requiring treatment of inhaled or systemic corticosteroids and/or routine use of beta-agonists or any controller drugs
* Use of antibiotic therapy for acute conditions within 14 days preceding the Screening Visit
* Exposure to systemic corticosteroids for any indication, chronic or intermittent within 60 days preceding the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2006-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Onset of action, measured by change from baseline in Total Nasal Symptom Score.

SECONDARY OUTCOMES:
changes in symptoms, safety.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Altana Pharma/Nycomed, Ontario, Mississauga, Canada

REFERENCES:
- See also: BY9010-M1-413-RDS-2007-06-05.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4538&filename=BY9010-M1-413-RDS-2007-06-05.pdf